CLINICAL TRIAL: NCT02316808
Title: Cholesterol-lowering Effects of Plant Stanol Ester
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Raisio Group (Industry)
Collaborators: Indonesia University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PCL_2011_Kal
Record Dates: First submitted 2014-12-10; First posted 2014-12-15 (Estimated); Last update posted 2014-12-23 (Estimated); Status verified 2014-12

CONDITIONS: Dyslipidemias; Hypercholesterolemia; Hyperlipidemias
MeSH Terms: conditions — Dyslipidemias; Hypercholesterolemia; Hyperlipidemias | interventions — plant stanol ester

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Placebo smoothie (Placebo Comparator)
  Interventions: Dietary Supplement: placebo
- Plant stanol ester smoothie (Experimental)
  Interventions: Dietary Supplement: Plant stanol ester

INTERVENTIONS:
Dietary Supplement: Plant stanol ester — Smoothie that contains plant stanol ester
  Arms: Plant stanol ester smoothie
Dietary Supplement: placebo — Smoothie that contains placebo
  Arms: Placebo smoothie

SUMMARY:
Efficacy of plant stanols as esters on LDL-cholesterol reduction is well documented. LDL-cholesterol lowering efficacy of the ingredient administered in a smoothie is less well known.

ELIGIBILITY:
Inclusion Criteria:

* total cholesterol concentration ≥ 200 mg/dL and < 300 mg/dL, and or LDL-C concentration ≥ 130 mg/dL and < 180 mg/dL
* were willing to consume control or plant stanol ester smoothie drinks two bottles per day immediately after a meal for four weeks,
* reachable by phone
* willing to declare written informed consent
* agreed in accordance with data protective stipulations and readiness to participate in the trial and to adhere to the study conditions.

Exclusion Criteria:

* Pregnant women
* obese
* diabetic subjects or subjects with random plasma glucose concentration > 200 mg/dL
* hyperthyroidism, a history of metabolic, endocrine and kidney disorders
* acute or chronic severe diseases possibly interfering with the evaluation of the outcome of the clinical trial (such as AIDS, tumor diseases, malignant hypertension, cardiac insufficiency according to NYHA III-IV)
* taking lipid-lowering medication or other medications likely to affect lipid metabolism

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2011-08; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Change (proportional) in LDL-C from baseline up to 4-weeks after plant stanol ester smoothie drink consumption. | 4 weeks

REFERENCES:
- [Derived] Lestiani L, Chandra DN, Laitinen K, Ambarwati FD, Kuusisto P, Lukito W. Double-Blind Randomized Placebo Controlled Trial Demonstrating Serum Cholesterol Lowering Efficacy of a Smoothie Drink with Added Plant Stanol Esters in an Indonesian Population. Cholesterol. 2018 Feb 4;2018:4857473. doi: 10.1155/2018/4857473. eCollection 2018. PMID 29535869